CLINICAL TRIAL: NCT05204277
Title: Clinical Evaluation of Different Minimal Invasive Treatment Modalities of Mild to Moderate Dental Fluorosis Using an Intra-oral Spectrophotometer
Brief Title: Clinical Evaluation of Dental Fluororsis Treatment Modalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Mostafa Nasser Abdelmoniem Youssef, Mostafa Nasser Abdelmoniem Youssef, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #202/2019
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Dental Fluorosis
Keywords: Bleaching, microabrasion, CPP-ACFP, color change, ∆E
MeSH Terms: conditions — Fluorosis, Dental | interventions — opalustre

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Masking was ensured as the baseline and follow-ups data were stored on a computer with a unique ID and the investigators were not disclosed about the participants' treatment protocol. Blinding of the participants was guaranteed as they didn't know each other, or the treatments received in other protocols
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- In-office bleaching (Active Comparator): 40% hydrogen peroxide in-office bleaching (Opalescence™ boost™ PF 40%, Ultradent Products, Inc., South Jordan, UT, USA)
  Interventions: Other: Opalescence™ boost™ PF 40%
- microabrasion (Active Comparator): 6.6% hydrochloric acid and silicon carbide microparticles microabrasion paste (Opalustre™, Ultradent Products, Inc., South Jordan, UT, USA)
  Interventions: Other: Opalustre™
- Remineralization (Active Comparator): casein phosphopeptide amorphous calcium fluoride phosphate (CPP-ACFP) remineralizing tooth crème (MI-Paste Plus®, GC America Inc., USA).
  Interventions: Other: MI-Paste Plus®
- Microabrasion + In-office bleaching (Active Comparator): teeth were treated with enamel microabrasion followed by in-office bleaching.
  Interventions: Other: Opalescence™ boost™ PF 40%; Other: Opalustre™
- In-office bleaching + Remineralization (Active Comparator): In-office bleaching was applied followed by MI-Paste Plus®
  Interventions: Other: Opalescence™ boost™ PF 40%; Other: MI-Paste Plus®
- Microabrasion + Remineralization (Active Comparator): microabrasion was applied followed by MI-Paste Plus®
  Interventions: Other: Opalustre™; Other: MI-Paste Plus®
- Microabrasion + In-office bleaching + Remineralization (Active Comparator): teeth were treated with microabrasion followed by inoffice bleaching and lastly MI-Paste Plus®
  Interventions: Other: Opalescence™ boost™ PF 40%; Other: Opalustre™; Other: MI-Paste Plus®
- Control (No Intervention): no treatment (control)

INTERVENTIONS:
Other: Opalescence™ boost™ PF 40% — 40% hydrogen peroxide in-office bleaching
  Arms: In-office bleaching; In-office bleaching + Remineralization; Microabrasion + In-office bleaching; Microabrasion + In-office bleaching + Remineralization
Other: Opalustre™ — 6.6% hydrochloric acid and silicon carbide microparticles microabrasion paste
  Arms: Microabrasion + In-office bleaching; Microabrasion + In-office bleaching + Remineralization; Microabrasion + Remineralization; microabrasion
Other: MI-Paste Plus® — casein phosphopeptide amorphous calcium fluoride phosphate (CPP-ACFP) remineralizing tooth crème
  Arms: In-office bleaching + Remineralization; Microabrasion + In-office bleaching + Remineralization; Microabrasion + Remineralization; Remineralization

SUMMARY:
Background: Various treatment modalities are available to improve esthetics of fluorosed teeth based on its severity.

Aim: evaluate the clinical performance of different minimal invasive treatment protocols on mild to moderate fluorosed teeth.

Materials and Methods: Participants were randomly allocated in eight treatment protocols with twenty teeth (n=20) included in each protocol. (P1) Opalescence boost PF 40%. (P2) Opalustre. (P3) MI-Paste Plus. In (P4) teeth were treated with Opalustre + Opalescence boost PF 40%. In (P5) Opalescence boost PF 40% + MI-Paste Plus, while in (P6) Opalustre +MI-Paste Plus. Whereas (P7) Opalustre + Opalescence boost PF 40% + MI-Paste Plus. (P8) control. All teeth were evaluated for color change (∆E) immediately after treatment (T1), after 14 days (T2), after 3 months (T3) and after 6 months (T4).

Statistical analysis: Two-way ANOVA was applied to test the interaction between different variables. ANOVA repeated measures were followed by Duncan multiple range tests (DMRTs) to compare between groups.

DETAILED DESCRIPTION:
This study was conducted for clinical evaluation of the quality of different minimal-invasive treatment modalities and combination treatments in esthetics improvement of mild to moderate fluorosed teeth using two different evaluation methods.

Materials and Methods:

Materials used in this study were Opalustre™ (microabrasion paste of 6.6% hydrochloric acid and Silicon Carbide), Opalescence™ Boost™ PF 40% (in-office bleaching of 40% hydrogen peroxide) and MI-Paste Plus® (topical remineralizing tooth crème of casein phosphopeptide amorphous calcium fluoride phosphate).

One hundred and sixty fluorosed teeth were included in this study. Prior to the interventions, tooth color coordinates were clinically recorded by VITA Easyshade V based on CIE Lab color system as baseline records. After that teeth were randomly allocated in eight treatment protocols with twenty teeth (n=20) included in each protocol. Protocol one (P1) Opalescence™ boost™ PF 40%. Protocol two (P2) Opalustre™. Protocol three (P3) MI-Paste Plus®. In protocol four (P4) teeth were treated with Opalustre™ followed by Opalescence™ boost™ PF 40%. In protocol five (P5) Opalescence™ boost™ PF 40% was applied followed by MI-Paste Plus®, while in protocol six (P6) Opalustre™ was applied followed by MI-Paste Plus®. Whereas protocol seven (P7) teeth were treated with Opalustre™ followed by Opalescence™ boost™ PF 40% and lastly MI-Paste Plus®. Protocol eight (P8) control.

All teeth were evaluated immediately after treatment (T1), after 14 days (T2), after 3 months (T3) and after 6 months (T4). Color change was calculated from the formula ∆E=√((∆〖L)〗^2+(∆〖a)〗^2+〖(∆b)〗^2 ) , where ∆L, ∆a and ∆b were the difference between readings mean values at different evaluating times from the baseline readings. Photographs were taken; immediately after application (T1), after 14 days (T2), after 3 months (T3) and after 6 months (T4).

Data were collected, checked, revised and organized in tables and figures using Microsoft Excel 2016. Data were checked for normality using Kolmogorov-Smirnov at 0.05. ∆L, ∆a, ∆b, and ∆E were normally distributed (p>0.05) i.e. parametric data, two-way ANOVA was applied to test the interaction between different variables. ANOVA repeated measures were followed by Duncan multiple range tests (DMRTs) to compare between groups.

ELIGIBILITY:
Inclusion Criteria:

* Each participant had at least 8 teeth with mild to moderate dental fluorosis score 1-4 according to Thylstrup and Fejerskov index.

  * Participants of age range 20-35 years old
  * Good oral and general health
  * Had no caries or restorations on the teeth to be treated
  * Ability to return for periodic recalls

Exclusion Criteria:

* Hypersensitive teeth
* Any fixed orthodontic appliance
* Current or previous use of bleaching agents
* A history of allergies to tooth whitening product
* Smoking habits
* Pregnant or lactating women

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Color change (∆E) | Six Months
  The color measurement was carried out 3 consecutive times with the same evaluator. At each time the obtained values were converted to the corresponding L, a and b values provided by the manufacturer and the mean of three measurements was taken. Color change was calculated from the formula ∆E=√((∆〖L)〗^2+(∆〖a)〗^2+〖(∆b)〗^2 ) ,

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Suez canal university, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No